CLINICAL TRIAL: NCT01090492
Title: A Phase 2a Randomized Double-blinded, Placebo And Active Controlled Two Cohort Two Doses Cross-over Multi-center Clinical Study To Assess Efficacy Of A Once Daily Administration Of A Phosphodiesterase 5 Inhibitor (Pf-00489791) For The Treatment Of Vasospasm In Primary And Secondary Raynaud's Phenomenon
Brief Title: PF-00489791 For The Treatment Of Raynaud's
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A7331010; EudraCT 2010-019009-40; 2010-019009-40 (EudraCT Number)
Record Dates: First submitted 2010-03-18; First posted 2010-03-22 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Raynaud's Disease; Peripheral Vascular Disease
Keywords: Raynaud's phenomenon; vasospasm; scleroderma; systemic sclerosis; CREST; phosphodiesterase inhibitor
MeSH Terms: conditions — Raynaud Disease; Peripheral Vascular Diseases; Scleroderma, Diffuse; Scleroderma, Systemic | interventions — PF-00489791

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Secondary Raynaud 4 mg dose (period 1) (Experimental)
  Interventions: Drug: PF-00489791
- Secondary Raynaud 4 mg dose (period 2) (Experimental)
  Interventions: Drug: PF-00489791
- Secondary Raynaud 20 mg dose (period 1) (Experimental)
  Interventions: Drug: PF-00489791
- Secondary Raynaud 20 mg dose (period 2) (Experimental)
  Interventions: Drug: PF-00489791
- Primary Raynaud 4 mg dose (period 1) (Experimental)
  Interventions: Drug: PF-00489791
- Primary Raynaud 4 mg dose (period 2) (Experimental)
  Interventions: Drug: PF-00489791
- Primary Raynaud 20 mg dose (period 1) (Experimental)
  Interventions: Drug: PF-00489791
- Primary Raynaud 20 mg dose (period 2) (Experimental)
  Interventions: Drug: PF-00489791

INTERVENTIONS:
Drug: PF-00489791 — Subjects with Secondary Raynaud's Phenomenon will receive PF-00489791 4 mg once a day for the first 4 week cross over period and then placebo once a day for the second 4 week cross over period
  Arms: Secondary Raynaud 4 mg dose (period 1)
Drug: PF-00489791 — Subjects with Secondary Raynaud's Phenomenon will receive placebo once a day for the first 4 week cross over period and then PF-00489791 4 mg once a day for the second 4 week cross over period
  Arms: Secondary Raynaud 4 mg dose (period 2)
Drug: PF-00489791 — Subjects with Secondary Raynaud's Phenomenon will receive PF-00489791 20 mg once a day for the first 4 week cross over period and then placebo once a day for the second 4 week cross over period
  Arms: Secondary Raynaud 20 mg dose (period 1)
Drug: PF-00489791 — Subjects with Secondary Raynaud's Phenomenon will receive placebo once a day for the first 4 week cross over period and then PF-00489791 20 mg once a day for the second 4 week cross over period
  Arms: Secondary Raynaud 20 mg dose (period 2)
Drug: PF-00489791 — Subjects with Primary Raynaud's Phenomenon will receive PF-00489791 4 mg once a day for the first 4 week cross over period and then placebo once a day for the second 4 week cross over period
  Arms: Primary Raynaud 4 mg dose (period 1)
Drug: PF-00489791 — Subjects with Primary Raynaud's Phenomenon will receive placebo once a day for the first 4 week cross over period and then PF-00489791 4 mg once a day for the second 4 week cross over period
  Arms: Primary Raynaud 4 mg dose (period 2)
Drug: PF-00489791 — Subjects with Primary Raynaud's Phenomenon will receive PF-00489791 20 mg once a day for the first 4 week cross over period and then placebo once a day for the second 4 week cross over period
  Arms: Primary Raynaud 20 mg dose (period 1)
Drug: PF-00489791 — Subjects with Primary Raynaud's Phenomenon will receive placebo once a day for the first 4 week cross over period and then PF-00489791 20 mg once a day for the second 4 week cross over period
  Arms: Primary Raynaud 20 mg dose (period 2)

SUMMARY:
The investigators propose that once daily administration of PF-00489791, a phosphodiesterase inhibitor, will reduce vasospasm and improve symptoms and signs associated with Primary and Secondary Raynaud's Phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Active Raynaud's Phenomenon
* Stable disease and medication requirements over the previous two months
* For Secondary Raynaud's Phenomenon subjects, a diagnosis of scleroderma using the American College of Rheumatology criteria or by the presence of at least 3/5 features of CREST syndrome
* both sexes

Exclusion Criteria:

* Uncontrolled hypertension, diabetes mellitus, angina, or using oral nitrates
* Smoking within 3 months or smoking cessation using nicotine products
* Subjects currently taking sildenafil, tadalafil or vardenafil
* Subjects with ulnar arterial occlusive disease as shown by a modified Allen test
* Pregnant or breast feeding or considering pregnancy in next 4 months
* Participation in trial for investigational drug within 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2010-08-04 (Actual); Primary Completion 2011-05-31 (Actual); Study Completion 2011-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (55):
- United States (23):
  - Stanford Hospital and Outpatient Center, Redwood City, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Arthritis and Rheumatology of Georgia, Atlanta, Georgia
  - Rockford Orthopedic Associates, Rockford, Illinois
  - Diagnostic Rheumatology and Research, PC, Indianapolis, Indiana
  - Memorial Health System, Inc. dba Memorial Medical Group Clinical Research Institute, South Bend, Indiana
  - Johns Hopkins University - Division of Rheumatology, Baltimore, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - West Michigan Rheumatology, PLLC, Grand Rapids, Michigan
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - UMDNJ - Robert Wood Johnson Medical Center Clinical Research Center, New Brunswick, New Jersey
  - The Center for Rheumatology, Albany, New York
  - Regional Rheumatology Associates, Binghamton, New York
  - AAIR Research Center, Rochester, New York
  - East Penn Rheumatology Associates, PC, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Rheumatic Disease Associates, Ltd., Willow Grove, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas
  - Rainier Clinical Research Center, Inc., Renton, Washington
- Canada (4):
  - Arthritis Centre Health Sciences Centre, Winnipeg, Manitoba
  - St. Joseph's Health Centre, London, Ontario
  - Rheumatology Research Associates, Ottawa, Ontario
  - Sir Mortimer B. Davis, Jewish General Hospital, Montreal, Quebec
- Colombia (5):
  - Centro Integral de Reumatologia e Inmunologia CIREI, Bogota, Cundinamarca
  - Fundacion Instituto de Reumatologia Fernando Chalem, Bogota, Cundinamarca
  - Idearg Sas, Bogotá, Cundinamarca
  - Servimed E.U, Bucaramanga, Santander Department
  - Medicity S.A.S, Bucaramanga
- Czechia (3):
  - REVMATOLOGIE s.r.o.,, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Revmatologicky ustav, Prague
- Dermatologisches Ambulatorium Hamburg-Alstertal, Hamburg, Germany
- Hungary (3):
  - Semmelweis Egyetem, Ersebeszeti Klinika, Budapest
  - Bacs-Kiskun Megyei Onkormanyzat Korhaza Szegedi Tudomanyegyetem AOK Oktato Korhaza, Kecskemét
  - Vas Megyei Markusovszky Korhaz Nonprofit Zrt, Angiologiai Szakambulancia, Szombathely
- Mexico (3):
  - Unidad de Investigacion en Enfermedades Cronico Degenerativas, Guadalajara, Jalisco
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Hospital Angeles. Centro Medico del Potosi, San Luis Potosí City
- Poland (4):
  - Slaskie Centrum Osteoporozy, Katowice
  - Prywatna Praktyka Lekarska Dr Med. Pawel Hrycaj, Poznan
  - Prywatna Praktyka Lekarska Prof. UM Dr hab. med. Pawel Hrycaj, Poznan
  - Katedra i Klinika Dermatologii, Wenerologii i Alergologii Akademii Medycznej we Wroclawiu, Wroclaw
- South Korea (3):
  - Seoul National University Hospital, Rheumatology, Internal Medicine, Seoul
  - Yonsei University College of Medicine, Severance Hospital, Rheumatology, Internal Medicine, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital/ Rheumatology, Internal Medicine, Seoul
- Spain (3):
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Del Mar, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Sweden (3):
  - CTC, Centrum för klinisk provning, Sahlgrenska Universitetssjukhuset, Gothenburg
  - Reumatologkliniken Skanes Universitetssjukhus Lund, Lund
  - Karolinska Universitetssjukhuset Solna, Reumatologiska kliniken, Stockholm

REFERENCES:
- [Derived] Su KY, Sharma M, Kim HJ, Kaganov E, Hughes I, Abdeen MH, Ng JHK. Vasodilators for primary Raynaud's phenomenon. Cochrane Database Syst Rev. 2021 May 17;5(5):CD006687. doi: 10.1002/14651858.CD006687.pub4. PMID 33998674
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7331010&StudyName=PF-00489791%20For%20The%20Treatment%20Of%20Raynaud%27s

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 243 participants were stratified into 2 cohorts (Primary Raynaud's phenomenon[PRP] and secondary RP[SRP]), who entered a 2-week placebo run-in period (to establish baseline), followed by a cross-over period (first 4 week treatment period,then a 2 week placebo washout,then 4 week treatment period) and then a 2-week placebo run-out period.
Groups:
- PRP Cohort: Placebo First, Then PF-00489791 4 mg: Two placebo tablets matched to PF-00489791 orally once daily for 4 weeks in first intervention period and then PF-00489791 tablets 4 milligram (mg) (2 tablets of PF-00489791 2 mg) orally once daily for 4 weeks in second intervention period to participants with PRP. A washout period of 2 weeks was maintained between each intervention period during which 2 placebo tablets matched to PF-00489791 were given orally once daily.
- PRP Cohort: PF-00489791 4mg First, Then Placebo: PF-00489791 tablets 4 mg (2 tablets of PF-00489791 2 mg) orally once daily for 4 weeks in first intervention period and then 2 placebo tablets matched to PF-00489791 orally once daily for 4 weeks in second intervention period to participants with PRP. A washout period of 2 weeks was maintained between each intervention period during which 2 placebo tablets matched to PF-00489791 were given orally once daily.
- PRP Cohort: Placebo First, Then PF-00489791 20 mg: Two placebo tablets matched to PF-00489791 orally once daily for 4 weeks in first intervention period and then PF-00489791 tablets 20 mg (2 tablets of PF-00489791 10 mg) orally once daily for 4 weeks in second intervention period to participants with PRP. A washout period of 2 weeks was maintained between each intervention period during which 2 placebo tablets matched to PF-00489791 were given orally once daily.
- PRP Cohort: PF-00489791 20 mg First, Then Placebo: PF-00489791 tablets 20 mg (2 tablets of PF-00489791 10 mg) orally once daily for 4 weeks in first intervention period and then 2 placebo tablets matched to PF-00489791 orally once daily for 4 weeks in second intervention period to participants with PRP. A washout period of 2 weeks was maintained between each intervention period during which 2 placebo tablets matched to PF-00489791 were given orally once daily.
- SRP Cohort: Placebo First, Then PF-00489791 4 mg: Two placebo tablets matched to PF-00489791 orally once daily for 4 weeks in first intervention period and then PF-00489791 tablets 4 milligram (mg) (2 tablets of PF-00489791 2 mg) orally once daily for 4 weeks in second intervention period to participants with SRP. A washout period of 2 weeks was maintained between each intervention period during which 2 placebo tablets matched to PF-00489791 were given orally once daily.
- SRP Cohort: PF-00489791 4 mg First, Then Placebo: PF-00489791 tablets 4 mg (2 tablets of PF-00489791 2 mg) orally once daily for 4 weeks in first intervention period and then 2 placebo tablets matched to PF-00489791 orally once daily for 4 weeks in second intervention period to participants with SRP. A washout period of 2 weeks was maintained between each intervention period during which 2 placebo tablets matched to PF-00489791 were given orally once daily.
- SRP Cohort: Placebo First, Then PF-00489791 20 mg: Two placebo tablets matched to PF-00489791 orally once daily for 4 weeks in first intervention period and then PF-00489791 tablets 20 mg (2 tablets of PF-00489791 10 mg) orally once daily for 4 weeks in second intervention period to participants with SRP. A washout period of 2 weeks was maintained between each intervention period during which 2 placebo tablets matched to PF-00489791 were given orally once daily.
- SRP Cohort: PF-00489791 20 mg First, Then Placebo: PF-00489791 tablets 20 mg (2 tablets of PF-00489791 10 mg) orally once daily for 4 weeks in first intervention period and then 2 placebo tablets matched to PF-00489791 orally once daily for 4 weeks in second intervention period to participants with SRP. A washout period of 2 weeks was maintained between each intervention period during which 2 placebo tablets matched to PF-00489791 were given orally once daily.
Period: First Intervention Period (4 Weeks)
Arm/Group | PRP Cohort: Placebo First, Then PF-00489791 4 mg | PRP Cohort: PF-00489791 4mg First, Then Placebo | PRP Cohort: Placebo First, Then PF-00489791 20 mg | PRP Cohort: PF-00489791 20 mg First, Then Placebo | SRP Cohort: Placebo First, Then PF-00489791 4 mg | SRP Cohort: PF-00489791 4 mg First, Then Placebo | SRP Cohort: Placebo First, Then PF-00489791 20 mg | SRP Cohort: PF-00489791 20 mg First, Then Placebo
Started | 27 | 29 | 29 | 28 | 33 | 32 | 32 | 33
Completed | 26 | 24 | 26 | 22 | 29 | 30 | 31 | 27
Not Completed | 1 | 5 | 3 | 6 | 4 | 2 | 1 | 6
Not completed — Protocol Violation | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0
Not completed — Did not meet inclusion criteria | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 3 | 1 | 2 | 0 | 5
Period: Placebo Washout Period ( 2 Weeks)
Arm/Group | PRP Cohort: Placebo First, Then PF-00489791 4 mg | PRP Cohort: PF-00489791 4mg First, Then Placebo | PRP Cohort: Placebo First, Then PF-00489791 20 mg | PRP Cohort: PF-00489791 20 mg First, Then Placebo | SRP Cohort: Placebo First, Then PF-00489791 4 mg | SRP Cohort: PF-00489791 4 mg First, Then Placebo | SRP Cohort: Placebo First, Then PF-00489791 20 mg | SRP Cohort: PF-00489791 20 mg First, Then Placebo
Started | 26 | 24 | 26 | 22 | 29 | 30 | 31 | 27
Completed | 26 | 24 | 26 | 22 | 29 | 30 | 31 | 27
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention Period (4 Weeks)
Arm/Group | PRP Cohort: Placebo First, Then PF-00489791 4 mg | PRP Cohort: PF-00489791 4mg First, Then Placebo | PRP Cohort: Placebo First, Then PF-00489791 20 mg | PRP Cohort: PF-00489791 20 mg First, Then Placebo | SRP Cohort: Placebo First, Then PF-00489791 4 mg | SRP Cohort: PF-00489791 4 mg First, Then Placebo | SRP Cohort: Placebo First, Then PF-00489791 20 mg | SRP Cohort: PF-00489791 20 mg First, Then Placebo
Started | 26 | 24 | 26 | 22 | 29 | 30 | 31 | 27
Completed | 25 | 22 | 24 | 22 | 27 | 29 | 22 | 25
Not Completed | 1 | 2 | 2 | 0 | 2 | 1 | 9 | 2
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Non-compliance | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 1 | 7 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- PRP Cohort: PF-00489791 4mg First, Then Placebo: PF-00489791 tablets 4 mg (2 tablets of PF-00489791 2 mg) orally once daily for 4 weeks in first intervention DB period and 2 placebo tablets matched to PF-00489791 orally once daily for 4 weeks in second DB intervention period to participants with PRP. A washout period of 2 weeks was maintained between each intervention period during which 2 placebo tablets matched to PF-00489791 were given orally once daily.
- PRP Cohort: Placebo First, Then PF-00489791 20 mg: Two placebo tablets matched to PF-00489791 orally once daily for 4 weeks in first intervention period and then PF-00489791 tablets 20 mg (2 tablets of PF-00489791 10 mg) orally once daily for 4 weeks in second DB intervention period to participants with PRP. A washout period of 2 weeks was maintained between each intervention period during which 2 placebo tablets matched to PF-00489791 were given orally once daily.
- Total: Total of all reporting groups
Arm/Group | PRP Cohort: Placebo First, Then PF-00489791 4 mg | PRP Cohort: PF-00489791 4mg First, Then Placebo | PRP Cohort: Placebo First, Then PF-00489791 20 mg | PRP Cohort: PF-00489791 20 mg First, Then Placebo | SRP Cohort: Placebo First, Then PF-00489791 4 mg | SRP Cohort: PF-00489791 4 mg First, Then Placebo | SRP Cohort: Placebo First, Then PF-00489791 20 mg | SRP Cohort: PF-00489791 20 mg First, Then Placebo | Total
Number analyzed (Participants) | 27 | 29 | 29 | 28 | 33 | 32 | 32 | 33 | 243
Age, Customized [Count of Participants; unit: Participants]
  Between 18 to 44 years | 14 | 12 | 14 | 14 | 10 | 6 | 16 | 9 | 95
  Between 45 to 64 years | 13 | 16 | 15 | 14 | 22 | 26 | 16 | 24 | 146
  Greater than or equal to (>=) 65 years | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 25 | 26 | 30 | 30 | 31 | 28 | 220
  Male | 2 | 4 | 4 | 2 | 3 | 2 | 1 | 5 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Raynaud's Condition Score (RCS) at Week 4
Description: The Raynaud's Condition score (RCS) is participant's rating of difficulty considering number of attacks, duration, amount of pain, numbness, or other symptoms caused in the fingers (including painful sores) due to the Raynaud's phenomenon every day and impact of Raynaud's alone on use of hands every day. An 11 point Likert scale is used to rate the difficulty caused by the condition each day with 0 = no difficulty and 10 = extreme difficulty. Participants were asked to select the number that best describes their difficulty, with higher score indicating worse condition. Average daily score was considered for participants completing more than 1 Raynaud's pain score scale on a day. Baseline value was calculated as mean of the scores over 7 days prior to treatment start. Week 4 value was calculated as mean of the scores over the 7-day period prior to Week 4.
Time Frame: Baseline, Week 4
Population: Per-protocol analysis set (PPAS) included all randomized participants compliant with diary completion and were not amongst serious protocol violators, receiving study medication till the study completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PF-00489791 4 mg (PRP): PF-00489791 tablets 4 mg (2 tablets of PF-00489791 2 mg) orally once daily for 4 weeks in first or second intervention period to participants with PRP.
- PF-00489791 20 mg (PRP): PF-00489791 tablets 20 mg (2 tablets of PF-00489791 10 mg) orally once daily for 4 weeks in first or second intervention period to participants with PRP.
- Placebo (PRP): Two placebo tablets matched to PF-00489791 orally once daily for 4 weeks in first or second intervention period to participants with PRP.
- PF-00489791 4 mg (SRP): PF-00489791 tablets 4 mg (2 tablets of PF-00489791 2 mg) orally once daily for 4 weeks in first or second intervention period to participants with SRP.
- PF-00489791 20 mg (SRP): PF-00489791 tablets 20 mg (2 tablets of PF-00489791 10 mg) orally once daily for 4 weeks in first or second intervention period to participants with SRP.
- Placebo (SRP): Two placebo tablets matched to PF-00489791 orally once daily for 4 weeks in first or second intervention period to participants with SRP.
Arm/Group | PF-00489791 4 mg (PRP) | PF-00489791 20 mg (PRP) | Placebo (PRP) | PF-00489791 4 mg (SRP) | PF-00489791 20 mg (SRP) | Placebo (SRP)
Number analyzed (Participants) | 34 | 39 | 73 | 47 | 36 | 83
units on a scale
  Baseline | 3.04 (1.899) | 2.90 (2.160) | 2.98 (1.958) | 3.14 (2.431) | 2.53 (1.833) | 2.97 (2.492)
  Change at Week 4 | -0.76 (1.901) | -1.05 (1.771) | -0.61 (1.404) | -0.82 (1.624) | -0.15 (1.090) | -0.24 (1.437)
Statistical Analysis 1: Comparison: PF-00489791 4 mg (PRP) vs Placebo (PRP); PRP: Adjusted mean difference analysis was based on Analysis of Covariance (ANCOVA) model with sequence, period and treatment as fixed effects and participant within sequence as a random effect, utilizing the baseline scores as covariate; Test type: Superiority or Other; p = 0.6513, ANCOVA; Adjusted Mean Difference = 0.11, 80% CI 2-sided [-0.21 to 0.44]
Statistical Analysis 2: Comparison: PF-00489791 20 mg (PRP) vs Placebo (PRP); PRP: Adjusted mean difference analysis was based on ANCOVA model with sequence, period and treatment as fixed effects and participant within sequence as a random effect, utilizing the baseline scores as covariate; Test type: Superiority or Other; p = 0.0057, ANCOVA; Adjusted Mean Difference = -0.69, 80% CI 2-sided [-0.99 to -0.38]
Statistical Analysis 3: Comparison: PF-00489791 4 mg (SRP) vs Placebo (SRP); SRP: Adjusted mean difference analysis was based on ANCOVA model with sequence, period and treatment as fixed effects and participant within sequence as a random effect, utilizing the baseline scores as covariate; Test type: Superiority or Other; p = 0.1157, ANCOVA; Adjusted Mean Difference = -0.44, 80% CI 2-sided [-0.80 to -0.08]
Statistical Analysis 4: Comparison: PF-00489791 20 mg (SRP) vs Placebo (SRP); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.6286, ANCOVA; Adjusted Mean Difference = -0.15, 80% CI 2-sided [-0.56 to 0.25]

2. Secondary Outcome: Change From Baseline in the Number of Raynaud's Attacks at Week 1, 2, 3 and 4
Description: Change from baseline in the number of Raynaud's attacks at Week 1, Week 2, Week 3 and Week 4 was calculated from the number of attacks reported over the 7-day period prior to each week from the patient diary, respectively.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4
Population: PPAS included all randomized participants compliant with diary completion and were not amongst serious protocol violators, receiving study medication till the study completion. Here, number analyzed signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Raynaud's attacks
Arm/Group | PF-00489791 4 mg (PRP) | PF-00489791 20 mg (PRP) | Placebo (PRP) | PF-00489791 4 mg (SRP) | PF-00489791 20 mg (SRP) | Placebo (SRP)
Number analyzed (Participants) | 34 | 39 | 73 | 47 | 36 | 83
Raynaud's attacks
  Baseline | 22.06 (20.587) | 16.31 (10.885) | 20.19 (17.802) | 22.80 (16.270) | 23.70 (20.909) | 23.08 (20.698)
  Change at Week 1 | -3.75 (7.494) | -2.47 (6.477) | -1.41 (7.934) | -3.17 (7.994) | -4.49 (14.692) | -2.36 (11.850)
  Change at Week 2 | -5.30 (9.487) | -2.36 (8.371) | -2.45 (11.107) | -3.76 (9.028) | -4.43 (17.312) | -1.87 (11.051)
  Change at Week 3 | -4.66 (10.559) | -4.86 (5.681) | -4.03 (10.396) | -4.25 (11.408) | -3.75 (8.601) | -1.93 (9.487)
  Change at Week 4: number analyzed (Participants) | 34 | 39 | 73 | 47 | 36 | 82
  Change at Week 4 | -4.85 (13.008) | -3.07 (7.118) | -3.65 (10.460) | -3.89 (8.326) | -2.68 (10.002) | -2.25 (10.624)
Statistical Analysis 1: Comparison: PF-00489791 4 mg (PRP) vs Placebo (PRP); At Week 4 - PRP: Adjusted mean difference analysis was based on ANCOVA model with sequence, period and treatment as fixed effects and participant within sequence as a random effect, utilizing the baseline scores as covariate; Test type: Superiority or Other; p = 0.9504, ANCOVA; Adjusted Mean Difference = 0.12, 80% CI 2-sided [-2.43 to 2.68]
Statistical Analysis 2: Comparison: PF-00489791 20 mg (PRP) vs Placebo (PRP); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4651, ANCOVA; Adjusted Mean Difference = -1.35, 80% CI 2-sided [-3.74 to 1.03]
Statistical Analysis 3: Comparison: PF-00489791 4 mg (SRP) vs Placebo (SRP); At Week 4 - SRP: Adjusted mean difference analysis was based on ANCOVA model with sequence, period and treatment as fixed effects and participant within sequence as a random effect, utilizing the baseline scores as covariate; Test type: Superiority or Other; p = 0.7423, ANCOVA; Adjusted Mean Difference = -0.59, 80% CI 2-sided [-2.92 to 1.73]
Statistical Analysis 4: Comparison: PF-00489791 20 mg (SRP) vs Placebo (SRP); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.3524, ANCOVA; Adjusted Mean Difference = -1.91, 80% CI 2-sided [-4.55 to 0.73]

3. Secondary Outcome: Change From Baseline in Mean Duration of Raynaud's Attacks at Week 4
Description: Mean duration of Raynaud's attacks for a time period was calculated as sum of recorded durations of attacks in the time period divided by total number of attacks in the time period where duration was recorded.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes per attack
Arm/Group | PF-00489791 4 mg (PRP) | PF-00489791 20 mg (PRP) | Placebo (PRP) | PF-00489791 4 mg (SRP) | PF-00489791 20 mg (SRP) | Placebo (SRP)
Number analyzed (Participants) | 34 | 39 | 73 | 47 | 36 | 83
minutes per attack
  Baseline | 17.69 (13.184) | 22.23 (36.562) | 19.61 (40.603) | 19.37 (18.929) | 19.07 (18.196) | 19.91 (19.886)
  Change at Week 4: number analyzed (Participants) | 34 | 39 | 73 | 47 | 36 | 82
  Change at Week 4 | -2.89 (7.480) | -5.63 (43.067) | -1.41 (12.348) | -3.92 (11.336) | -2.61 (9.593) | -1.65 (10.609)
Statistical Analysis 1: Comparison: PF-00489791 4 mg (PRP) vs Placebo (PRP); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.7900, ANCOVA; Adjusted Mean Difference = 1.21, 80% CI 2-sided [-4.61 to 7.03]
Statistical Analysis 2: Comparison: PF-00489791 20 mg (PRP) vs Placebo (PRP); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1463, ANCOVA; Adjusted Mean Difference = -6.17, 80% CI 2-sided [-11.61 to -0.73]
Statistical Analysis 3: Comparison: PF-00489791 4 mg (SRP) vs Placebo (SRP); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.1446, ANCOVA; Adjusted Mean Difference = -2.37, 80% CI 2-sided [-4.44 to -0.29]
Statistical Analysis 4: Comparison: PF-00489791 20 mg (SRP) vs Placebo (SRP); [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.5497, ANCOVA; Adjusted Mean Difference = -1.09, 80% CI 2-sided [-3.45 to 1.26]

4. Secondary Outcome: Change From Baseline in the Mean Raynaud's Pain Score at Week 1, 2, 3 and 4
Description: Participants were asked to rate their worst Raynaud's pain in the past 24 hours using an 11 point Likert scale, with 0 = no Raynaud's pain and 10 = the worst possible pain. Highest (most severe) response was considered for participants responding at more than 1 point on the scale. Average daily score was considered for participants completing more than 1 Raynaud's pain score scale on a day. Baseline value was calculated as mean of the scores over 7 days prior to treatment start. Post-baseline value was calculated as mean of the scores over the 7-day period prior to the visit.
Time Frame: Baseline, Week 1, 2, 3, 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-00489791 4 mg (PRP) | PF-00489791 20 mg (PRP) | Placebo (PRP) | PF-00489791 4 mg (SRP) | PF-00489791 20 mg (SRP) | Placebo (SRP)
Number analyzed (Participants) | 34 | 39 | 73 | 47 | 36 | 83
units on a scale
  Baseline | 2.84 (2.074) | 2.78 (2.348) | 2.80 (2.064) | 3.33 (2.614) | 2.54 (1.895) | 3.10 (2.753)
  Change at Week 1 | -0.72 (1.525) | -0.74 (1.266) | -0.26 (1.205) | -0.53 (1.440) | -0.32 (1.276) | -0.17 (1.272)
  Change at Week 2 | -0.94 (1.745) | -0.61 (1.524) | -0.48 (1.337) | -0.68 (1.740) | -0.33 (1.321) | -0.24 (1.306)
  Change at Week 3 | -0.82 (1.720) | -1.12 (1.664) | -0.62 (1.262) | -0.80 (1.836) | -0.55 (1.081) | -0.33 (1.269)
  Change at Week 4: number analyzed (Participants) | 34 | 39 | 73 | 47 | 36 | 82
  Change at Week 4 | -0.80 (1.842) | -1.14 (1.820) | -0.63 (1.423) | -0.77 (1.922) | -0.35 (1.115) | -0.27 (1.466)
Statistical Analysis 1: Comparison: PF-00489791 4 mg (PRP) vs Placebo (PRP); Week 4 (PRP): Adjusted mean difference analysis was based on ANCOVA model with sequence, period and treatment as fixed effects and participant within sequence as a random effect, utilizing the baseline scores as covariate; Test type: Superiority or Other; p = 0.5909, ANCOVA; Adjusted Mean Difference = 0.15, 80% CI 2-sided [-0.21 to 0.52]
Statistical Analysis 2: Comparison: PF-00489791 20 mg (PRP) vs Placebo (PRP); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0053, ANCOVA; Adjusted Mean Difference = -0.77, 80% CI 2-sided [-1.12 to -0.43]
Statistical Analysis 3: Comparison: PF-00489791 4 mg (SRP) vs Placebo (SRP); Week 4 (SRP): Adjusted mean difference analysis was based on ANCOVA model with sequence, period and treatment as fixed effects and participant within sequence as a random effect, utilizing the baseline scores as covariate; Test type: Superiority or Other; p = 0.3462, ANCOVA; Adjusted Mean Difference = -0.28, 80% CI 2-sided [-0.67 to 0.10]
Statistical Analysis 4: Comparison: PF-00489791 20 mg (SRP) vs Placebo (SRP); [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.1940, ANCOVA; Adjusted Mean Difference = -0.44, 80% CI 2-sided [-0.88 to -0.01]

5. Secondary Outcome: Number of Participants With Decrease From Baseline in Digital Ulcers at Day 14 and 28: Secondary Raynaud's Phenomenon Cohort
Description: Presence of ulcer was assessed at baseline. At post-baseline visits, each ulcer was measured and scored: 1= smaller or improved compared to previous visit, 2= same as previous visit, 3= bigger or worse than previous visit, and 4= new. If a new digital ulcer develops during the course of the study, the measurement and scoring were initiated on this additional ulcer. Healed ulcers were not counted into the number of ulcers. Participants with SRP in the per-protocol population with at least 1 digital ulcer present at any assessment were evaluable for this measure. Results are reported for participants with presence of ulcer at baseline and decrease from baseline in ulcers at post-baseline visits.
Time Frame: Baseline, Day 14, 28
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | PF-00489791 4 mg (SRP) | PF-00489791 20 mg (SRP) | Placebo (SRP)
Number analyzed (Participants) | 47 | 36 | 83
participants
  Baseline: number analyzed (Participants) | 47 | 36 | 79
  Baseline | 10 | 7 | 16
  With Decrease at Day 14: number analyzed (Participants) | 10 | 7 | 17
  With Decrease at Day 14 | 7 | 1 | 6
  With Decrease at Day 28: number analyzed (Participants) | 11 | 8 | 19
  With Decrease at Day 28 | 9 | 5 | 7

6. Secondary Outcome: Plasma Concentration of PF-00489791 and Its Metabolites
Description: Only participants receiving PF-00489791 were to be analyzed for this outcome. Data have been calculated by setting plasma concentration values below the lower limit of quantification to 0. The lower limit of quantification is 0.0100 microgram per milliliter (mcg/mL). Data for plasma concentration of PF-00489791 metabolites was not analyzed, as it was not intended to be a secondary endpoint and was deemed optional.
Time Frame: Day 1, 15, 29 (Day 1, 15, 29 for first intervention period), 43, 57, 71 (Day 1, 15, 29 for second intervention period)
Population: Analysis population included participants who received 1 dose of study drug and were analyzed for pharmacokinetic parameters. Here, Overall number of participants signifies participants evaluable for either first or second intervention period and number analyzed signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | PF-00489791 4 mg (PRP) | PF-00489791 20 mg (PRP) | PF-00489791 4 mg (SRP) | PF-00489791 20 mg (SRP)
Number analyzed (Participants) | 55 | 54 | 61 | 64
mcg/mL
  Day 1: number analyzed (Participants) | 29 | 28 | 32 | 33
  Day 1 | 0.0058 (0.0314) | NA (NA) — Number of observations above lower limit of quantification (NALQ) was 0, hence data could not be analyzed. | NA (NA) — Number of observations above lower limit of quantification (NALQ) was 0, hence data was not summarized. | NA (NA) — Number of observations above lower limit of quantification (NALQ) was 0, hence data was not summarized.
  Day 15: number analyzed (Participants) | 27 | 24 | 31 | 28
  Day 15 | 0.1523 (0.0855) | 0.5907 (0.3736) | 0.1756 (0.09038) | 0.7718 (0.4991)
  Day 29: number analyzed (Participants) | 24 | 22 | 31 | 28
  Day 29 | 0.1489 (0.0854) | 0.6525 (0.3822) | 0.1776 (0.08508) | 0.7577 (0.4137)
  Day 43: number analyzed (Participants) | 26 | 26 | 29 | 31
  Day 43 | NA (NA) — Number of observations above lower limit of quantification (NALQ) was 0, hence data could not be analyzed. | NA (NA) — Number of observations above lower limit of quantification (NALQ) was 0, hence data could not be analyzed. | NA (NA) — Number of observations above lower limit of quantification (NALQ) was 0, hence data was not summarized. | NA (NA) — Number of observations above lower limit of quantification (NALQ) was 0, hence data was not summarized.
  Day 57: number analyzed (Participants) | 25 | 24 | 27 | 22
  Day 57 | 0.1088 (0.0629) | 0.6890 (0.4318) | 0.1167 (0.05644) | 0.7565 (0.6224)
  Day 71: number analyzed (Participants) | 25 | 24 | 27 | 31
  Day 71 | 0.1178 (0.0614) | 0.6337 (0.3745) | 0.1224 (0.0638) | 0.6639 (0.5834)

7. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for laboratory tests abnormalities included: hemoglobin, hematocrit and red blood cells (less than [<] 0.8*lower limit of normal[LLN]); leukocytes (<0.6 LLN /greater than [>] 1.5*upper LN [ULN]; platelets (<0.5*LLN/>1.75*ULN); neutrophils, lymphocytes (<0.8* LLN/>1.2*ULN); eosinophils, basophils, monocytes (>1.2*ULN); bilirubin (>1.5*ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), Gamma GT, alkaline phosphatase (>3*ULN); BUN, creatinine (>1.3*ULN); glucose (<0.6 LLN/>1.5*ULN); uric acid (>1.2*ULN); sodium (<0.95*LLN/>1.05*ULN); potassium, calcium, chloride, bicarbonate (<0.9*LLN/>1.1*ULN); albumin, total protein (<0.8*LLN/>1.2*ULN); creatine kinase (>2.0*ULN); Urine Specific Gravity, Urine pH, urine blood, urine glucose, urine protein, urine ketones, urine leukocytes esterase (>=1 high-powered field). Total number of participants with any laboratory abnormalities was reported.
Time Frame: Screening up to 28 days after last study dose (up to 98 days)
Population: Analysis population included all randomized participants who took at least 1 dose of study medication along with at least 1 on-treatment laboratory test result.
Measure: Number; unit: participants
Arm/Group | PF-00489791 4 mg (PRP) | PF-00489791 20 mg (PRP) | Placebo (PRP) | PF-00489791 4 mg (SRP) | PF-00489791 20 mg (SRP) | Placebo (SRP)
Number analyzed (Participants) | 50 | 48 | 98 | 57 | 60 | 114
participants | 2 | 4 | 14 | 5 | 13 | 10

8. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs and Orthostatic Blood Pressure Measurements
Description: Vital signs assessment included measurement of supine and standing pulse rate, systolic and diastolic blood pressures. Criteria for clinically significant vital signs and orthostatic blood pressure measurements were based on investigator's judgement.
Time Frame: Screening up to 28 days after last study dose (up to 98 days)
Population: Safety analysis set consisted of all participants who took at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-00489791 4 mg (PRP) | PF-00489791 20 mg (PRP) | Placebo (PRP) | PF-00489791 4 mg (SRP) | PF-00489791 20 mg (SRP) | Placebo (SRP)
Number analyzed (Participants) | 55 | 54 | 102 | 61 | 64 | 122
participants | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Values
Description: ECG assessment included measurement of PR, QRS, QT,corrected QT interval (QTc)values. Criteria for clinically significant ECG values were based on investigator's judgement.
Time Frame: Screening up to 28 days after last study dose (up to 98 days)
Population: Safety analysis set consisted of all participants who took at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-00489791 4 mg (PRP) | PF-00489791 20 mg (PRP) | Placebo (PRP) | PF-00489791 4 mg (SRP) | PF-00489791 20 mg (SRP) | Placebo (SRP)
Number analyzed (Participants) | 55 | 54 | 102 | 61 | 64 | 122
participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Safety analysis population included all participants who received at least 1 dose of study medication.
Arm/Group | PF-00489791 4 mg (PRP) | PF-00489791 20 mg (PRP) | Placebo (PRP) | PF-00489791 4 mg (SRP) | PF-00489791 20 mg (SRP) | Placebo (SRP)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54 | 0/102 | 0/61 | 0/64 | 1/122
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54 | 0/102 | 0/61 | 0/64 | 1/122
Other Adverse Events (participants affected / at risk) | 27/55 | 34/54 | 43/102 | 34/61 | 51/64 | 60/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00489791 4 mg (PRP) (N=55) | PF-00489791 20 mg (PRP) (N=54) | Placebo (PRP) (N=102) | PF-00489791 4 mg (SRP) (N=61) | PF-00489791 20 mg (SRP) (N=64) | Placebo (SRP) (N=122)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00489791 4 mg (PRP) (N=55) | PF-00489791 20 mg (PRP) (N=54) | Placebo (PRP) (N=102) | PF-00489791 4 mg (SRP) (N=61) | PF-00489791 20 mg (SRP) (N=64) | Placebo (SRP) (N=122)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 2 | 2 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 4 | 0
Cystic fibrosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 1 | 1 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eye oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 4 | 0 | 7 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 5 | 0 | 2 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 3 | 2
Oesophageal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Salivary gland calculus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2 | 3
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 3 | 1 | 1 | 2
Feeling hot (General disorders) | 0 | 0 | 3 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 1 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 3 | 0
Oedema peripheral (General disorders) | 0 | 2 | 2 | 3 | 3 | 0
Pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 1 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alveolar osteitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 4
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 3 | 1 | 3 | 4
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 1 | 2 | 0 | 2 | 2
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 10 | 2 | 1 | 5
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Frostbite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2 | 5 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 4 | 7 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 0 | 2 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Benign neoplasm of cornea (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 3 | 3 | 4
Headache (Nervous system disorders) | 8 | 14 | 9 | 9 | 21 | 12
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Orgasm abnormal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erection increased (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Spontaneous penile erection (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acne cystic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 3 | 2 | 1 | 3 | 4 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Plasma concentration of PF-00489791 metabolites was not intended as secondary endpoint in the protocol and was considered as an exploratory endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.